CLINICAL TRIAL: NCT01329133
Title: Treatment of Severe and Resistant Obsessive-compulsive Disorder by High-frequency Stimulation of the Ventral Striatum and the Subthalamic Nucleus
Brief Title: Deep Brain Stimulation and Obsessive-compulsive Disorder
Acronym: STOC2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUBX 2010/43
Record Dates: First submitted 2011-04-04; First posted 2011-04-05 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Deep brain stimulation (DBS); Obsessive compulsive disorder; ventral striatum; subthalamic nucleus
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DBS of subthalamic nucleus (Active Comparator)
  Interventions: Procedure: Deep Brain Stimulation (DBS)
- DBS of ventral striatum (Active Comparator)
  Interventions: Procedure: Deep Brain Stimulation (DBS)

INTERVENTIONS:
Procedure: Deep Brain Stimulation (DBS) — In a first time: Implantation of DBS electrodes, stereotactically, in each hemisphere into the targeted brain structure under local anesthesia. In a second time (next week): installation of the deep brain neurostimulator and connection to the electrodes implanted under general anesthesia. And one month later: beginning of the stimulation.

SUMMARY:
Obsessive-compulsive disorder (OCD) is a relatively common psychiatric condition, which is classically treated by antidepressant medications in combination with psychotherapies. However, both these conventional therapeutic approaches fail to sufficiently improve obsessive-compulsive symptoms in 20-30% of cases. From these considerations, deep brain stimulation (DBS), as a reversible and adjustable surgical procedure, has recently been introduced in the field of resistant OCD. DBS currently uses electrodes with four contacts on each lead, which are bilaterally implanted into the chosen brain structure. DBS consists of the delivery of a high-frequency current through the quadripolar electrodes connected to a battery powered pulse-generating device. Several clinical investigations have shown that DBS, primarily targeting either the ventral striatum (VS) or the subthalamic nucleus (STN), as brain sites of interest because of their particular involvement in the production of OCD symptoms, is able to produce an approximately 40% or greater reduction in clinical symptom intensity in severely chronic and incapacitating forms of OCD. These promising findings lead to propose a comparison of the efficacy, safety and tolerability of DBS choosing either the VS or STN as brain target by conducting a large controlled trial and including a medico-economic analysis for assessing the classical cost/efficacy ratio. In this way, the present study is expected to promote and highlight the importance of DBS, as an effective, safe, well-tolerated and cost-relevant surgical approach for the management of resistant OCD.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a relatively common psychiatric condition with an estimated lifetime prevalence of 2-3 % of the general population. It is generally characterized by a chronic course leading to a profound impairment in psychosocial functioning and to a marked deterioration in quality of life. Today, the well-established efficacy of antidepressants, acting preferentially by blocking serotonin reuptake, in addition to psychological treatments, have considerably changed the poor prognosis of the illness. However, both conventional therapeutic approaches failed to substantially alleviate obsessive-compulsive symptoms in 20-30% of cases. Deep brain stimulation, as a reversible and adjustable surgical procedure, has recently been introduced in the field of OCD, primarily targeting either the ventral striatum (VS) or the subthalamic nucleus (STN) and leading to an approximately 40% or greater reduction in clinical symptom intensity from baseline levels in severely chronic and resistant forms of OCD. These promising findings lead to propose a comparison of the efficacy, safety and tolerability of DBS choosing either the VS or STN as brain target by conducting a multicenter, parallel-group, randomized, single-blind trial over a 13-month follow-up period. For this purpose, a total population of 28 OCD patients who meet the currently used operational criteria for defining therapeutic resistance will be recruited. The surgical procedure will consist in the implantation of stimulation electrodes with four contacts on each lead, which are stereotactically and bilaterally implanted into the targeted brain structure under local anesthesia. Per-operative, single-unit electrophysiological recordings of the neuronal activity will be performed using five parallel microelectrodes and serving as guide for the implantation of both definitive electrodes. They will be connected to a battery powered pulse-generating device five days later under general anesthesia. Thereafter, psychiatric assessments including both the Y-BOCS ("Yale-Brow Obsessive-compulsive scale") and PI ("Padua Inventory") for measuring OCD symptom severity, the BAS ("Brief Anxiety Scale"), MADRS ("Montgomery and Asberg Depression rating Scale") and HAD ("Hospital Anxiety and Depression Scale") for determining anxiety and/or depressive symptom intensity, and the CGI ("Clinical Global Impression") rating scales for evaluating global symptom severity and treatment response will be performed every 3 months beyond the one-month postoperative free-stimulation period. This will be coupled with a large battery of neuropsychological tests exploring all executive functions in combination with precise medical records of side effects for appreciating safety/tolerability of DBS. A cost-effectiveness analysis, as a formal method of comparing DBS and classical therapeutic strategies with regard to their respective resource utilization (costs) and outcomes (effectiveness) will also be carried out. Therefore, the present study may contribute to highlight the special interest of DBS, as an effective, safe, well-tolerated and cost-relevant surgical approach for the management of resistant OCD.

ELIGIBILITY:
Inclusion Criteria:

* Age comprised between 18 and 60 years
* History of OCD for at least 5 years according to the DSM-IV-TR criteria and characterized by a "good insight", as determined by the BABS ("Brown Assessment of Beliefs Scale")
* Severe form of OCD, as evidenced by:

  * a score ≥ 25 on the Y-BOCS
  * a score > 4 on the CGI scale
  * a score =< 40 on the GAF ("global assessment of functioning)
* Lack of therapeutic effects of at least 3 antidepressants selectively blocking serotonin reuptake (SSRI) at least 12 consecutive weeks at the maximal tolerated dose (up to 80 mg/day for fluoxetine, 300 mg/day for fluvoxamine, 200 mg/day for sertraline, 60 mg/day for paroxetine, 60mg/day for citalopram and 250 mg/day for clomipramine) prescribed alone and in combination for at least 1 month with: 1) risperidone or olanzapine or aripiprazole or quetiapine, 2) clomipramine
* Lack of therapeutic effects of behavioral therapy with two different therapists using conventional techniques primarily based on exposure with prevention of ritualized response
* Understand and accept the design and constraints of the present study
* Be a beneficiary or member of health insurance plan
* Provide written consent to the study after receiving clear information

Exclusion Criteria:

* Patient with cognitive impairment with a Mattis scale score ≤ 130
* Patient with other DSM-IV-TR axis I diagnoses (schizophrenia, bipolar, substance abuse or substance dependence), except for generalized anxiety disorder, social phobia or nicotine dependence
* Patient with high suicide risk, as indicated by a score ≥ 2 on the MADRS (item 10)
* Patient with personality disorder corresponding to the clusters A and B, as assessed with the SIDP-IV ("Structured Interview for DSM-IV Personality")
* Patient with contraindication for MRI scanning, abnormal brain MRI or serious intercurrent disease
* Patient with contraindication for surgery or anesthesia
* Patient currently treated with anticoagulant or antiplatelet drug
* Be a woman of childbearing age without effective contraception
* Be hospitalized under constraint
* Be under guardianship procedures
* Prohibition on participation in other research, apart from any other non-interventional research

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2011-04-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Combination of three criteria (composite criterion), as follows: a. Y-BOCS score ≤ 16 / and b. Technical feasibility (each leads in the target) / and c. Safety, as assessed by any serial adverse event | Month 13 : one year after stimulation

SECONDARY OUTCOMES:
Remission as defined by a Y-BOCS score ≤ 16 at M13 | Month 13 : one year after stimulation
Number of electrode contacts correctly located within the chosen brain target (0, 1 or 2) | End of surgical procedure (day 1)
Monitoring of psychological and somatic complaints made spontaneously by the patient over the course of the present trial, in combination to the semi-structured interview for collecting side effects | Every 3 months from Month 1 to Month 13
Scores on neuropsychological tests exploring all executive functions | Every 3 months from Month 1 to Month 13
Percentage change in the total Y-BOCS score from M1 to M13 | Every 3 months from Month 1 to Month 13
Therapeutic response, as indicated by a 35% decrease or more in the Y-BOCS score and a score of 1 or 2 (very much or much improved) on the CGI improvement scale from M1 to M13 | Every 3 months from Month 1 to Month 13
Percentage change in the Y-BOCS obsessive and compulsive subscores from M1 to M13 | Every 3 months from Month 1 to Month 13
Percentage change in the overall Padua Inventory score, MADRS score, BAS score from M1 to M13 | Every 3 months from Month 1 to Month 13
Percentage change in the total and depression and anxiety subscale scores on the HAD scale from M1 and M13 | Every 3 months from Month 1 to Month 13
Ratings of functional disability and quality of life | Every 3 months from Month 1 to Month 13
Correlations between efficacy and anatomical positioning of both stimulation electrodes within the chosen brain target | Every 3 months from Month 1 to Month 13
cost comparison of therapeutic strategies | M-13 and M13 (one year after stimultaion)
  cost comparison of thérapeutic strategies : classical versus surgical
Cost / effectiveness ration | M-13/ M13 (one year after stimulation)
  Cost / effectiveness ratio : cost difference between therapeutic strategies and success rate of DBS
Cost-utility rati | every 3 months from month 1 to month 13
  Cost-utility ratio based on SF-36 scores.

CONTACTS AND LOCATIONS:
Overall Officials: BENARD Antoine, MD, Study Chair — University Hospital Bordeaux, France; Emmanuel CUNY, MD, Principal Investigator — University Hospital Bordeaux, France; Bruno AOUIZERATE, MD-PhD, Principal Investigator — Charles Perrens hospital, Bordeaux, France
Locations (14):
- France (14):
  - Bordeaux University Hospital, Bordeaux
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Henri Mondor Hospital, Créteil
  - Grenoble University Hospital, Grenoble
  - Lille University Hospital, Lille
  - Lyon University Hospital, Lyon
  - Marseille University Hospital, Marseille
  - Nice University Hospital, Nice
  - Pitié-Salpêtrière Hospital, Paris
  - Sainte-Anne Hospital, Paris
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital, Rennes
  - Strasbourg University Hospital, Strasbourg
  - Toulouse University Hospital, Toulouse

REFERENCES:
- [Background] Aouizerate B, Cuny E, Bardinet E, Yelnik J, Martin-Guehl C, Rotge JY, Rougier A, Bioulac B, Tignol J, Mallet L, Burbaud P, Guehl D. Distinct striatal targets in treating obsessive-compulsive disorder and major depression. J Neurosurg. 2009 Oct;111(4):775-9. doi: 10.3171/2009.2.JNS0881. PMID 19284243
- [Background] Mallet L, Polosan M, Jaafari N, Baup N, Welter ML, Fontaine D, du Montcel ST, Yelnik J, Chereau I, Arbus C, Raoul S, Aouizerate B, Damier P, Chabardes S, Czernecki V, Ardouin C, Krebs MO, Bardinet E, Chaynes P, Burbaud P, Cornu P, Derost P, Bougerol T, Bataille B, Mattei V, Dormont D, Devaux B, Verin M, Houeto JL, Pollak P, Benabid AL, Agid Y, Krack P, Millet B, Pelissolo A; STOC Study Group. Subthalamic nucleus stimulation in severe obsessive-compulsive disorder. N Engl J Med. 2008 Nov 13;359(20):2121-34. doi: 10.1056/NEJMoa0708514. PMID 19005196